CLINICAL TRIAL: NCT04158856
Title: Adjuvant Dual Anti-HER2 Therapy in Patients With Tumors < 8mm, Node-negative, HER2-positive Breast Cancer :a Single-group Arm, Open-label, Prospective, Phase 2 Study
Brief Title: Adjuvant Dual Anti-HER2 Therapy in Patients With Small, Node-negative, HER2-positive Breast Cancer
Acronym: SHERO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: xuexin he (Other)
Responsible Party: Sponsor-Investigator, xuexin he, Associate chief physician, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHERO
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pyrotinib; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): adjuvant Pyrotinib plus Trastuzumab
  Interventions: Drug: Pyrotinib; Drug: Trastuzumab

INTERVENTIONS:
Drug: Pyrotinib — 400mg po every day
  Other Names: Pyrotinib Maleate Tablets
Drug: Trastuzumab — Trastuzumab is administered at a loading dose of 8 mg/kg IV followed by 6 mg/kg every 21 days
  Other Names: Herceptin

SUMMARY:
This phase II trial aims to study the efficacy and safety of adjuvant Pyrotinib plus trastuzumab in patients with tumors <8mm, node-negative, HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-70 years old
2. Have finished radical operation
3. Histologically confirmed invasive ductal carcinoma (IDCA)
4. According to AJCC ,pT<8mm, pN0, no evidence for metastasis
5. Operation specimens are available for ER, progesterone receptor (PR) and HER2 detection, patients should be HER2 positive tumor (IHC staining of 3+ [uniform, intense membrane staining of >30% of invasive tumor cells], or a FISH result of .6 HER2 gene copies per nucleus or a FISH ratio [HER2 gene signals to chromosome 17 signals] of >2.2), nuclear grade 3.
6. Should have tumor tissue available and sufficient for multi-spots sampling.
7. It has been <84 days since the date of definitive surgery, and there is adequate wound healing as determined by the Treating Physician.
8. Has Eastern Cooperative Oncology Group (ECOG) Performance Score 0-1, expected survival time > 12 months
9. Cardiac function had to be within normal limits (left ventricular ejection fraction [LVEF] ≥50%), as established by multiple gated acquisition scan or echocardiography.
10. Adequate bone marrow function, adequate liver and renal function, and adequate coagulation function.
11. Women with potential child-bearing must have a negative pregnancy test (urine or serum) within 7 days of drug administration and agree to use an acceptable and effective method of contraception to avoid pregnancy during the study.
12. Written informed consent according to the local ethics committee requirements.

Exclusion Criteria:

1. pT≥8mm or node positive
2. Metastatic breast cancer
3. Any prior systemic or loco-regional treatment of breast cancer, including chemotherapy in 28 days
4. With a history of malignant tumor except uterine cervix cancer in situ or skin basal cell carcinoma
5. Patients with medical conditions that indicate intolerant to adjuvant target therapy and related treatment, including severe infection, coagulation disorder, active peptic ulcer, coagulation disorder, connective tissue disease or myelo-suppressive disease
6. Has symptomatic peripheral neuropathy > grade 2 according to NCI
7. Known severe allergy to any drugs in this study
8. Has cardiac dysfunction or lung dysfunction defined as follows:

   * grade ≥3 CHF according to NCI CTCAE v 5.0 or NYHA≥II
   * angina which requires drug control, cardiac infraction, and any other vascular disease with apparent clinical symptoms
   * uncontrolled high-risk arrhythmia
   * uncontrolled hypertension
9. Has active hepatitis B or hepatitis C with abnormal liver function tests (LFTs) or is known to be HIV positive
10. Patient is pregnant or breast feeding

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | 5 years
  stimated percentage of patients alive and disease-free at 5 years from randomization or censored at date of last follow-up.

SECONDARY OUTCOMES:
Breast Cancer Specific Survival | 5 years
  Estimated percentage of patients alive and disease-free at 5 years from randomization, where breast cancer specific survival is defined as the time from randomization to death from breast cancer relapse; or censored at date last known alive.
Overall Survival | 5 years
  Estimated percentage of patients alive and disease-free at 5 years from randomization, where overall survival is defined as the time from randomization to death from any cause; or censored at date last known alive.
Treatment-related adverse events | up to 3 months
  Incidence and severity of adverse events as assessed by NCI CTCAE V5.0
Change of LVEF after treatment | up to 3 months
  The change of LVEF after 3 months treatment compared to the baseline LVEF

CONTACTS AND LOCATIONS:
Overall Officials: Xuexin He, MD, Study Chair — Seaond Affiliated Hospital, Zhejiang University, School of Medicine